CLINICAL TRIAL: NCT01414621
Title: IRB #14547: Expression of Angiogenic Factors in Myocardial Tissue in Diabetic and Non-diabetic Patients Undergoing Coronary Bypass Surgery
Brief Title: Expression of Angiogenic Factors in Myocardial Tissue
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jacob Raphael, Attending Anesthesiologist, University of Virginia
Other Study IDs: 14547
Record Dates: First submitted 2010-09-17; First posted 2011-08-11 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: CABG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the cannulation process before the initiation of CPB(cardiopulmonary bypass) a small piece of right atrial tissue is cut in order to insert venous drainage cannula to the right atrium. This small piece of tissue is discarded and is not sent for pathology.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG patients: atrial tissue samples from CABG patients
  Interventions: Other: atrial tissue sample

INTERVENTIONS:
Other: atrial tissue sample — atrial tissue sample from CABG patient

SUMMARY:
The purpose of this study is to evaluate whether angiogenesis is decreased in diabetic patients with coronary artery disease compared to non-diabetics with coronary artery disease. The protein expression of angiogenic factors will be examined in atrial tissue prior to initiation of cardiopulmonary bypass in patients undergoing coronary bypass surgery.

The goal of this project is to evaluate the tissue levels of HIF-1, VEGF and angiostatin in diabetic and non-diabetic patients coming for on-pump coronary artery bypass graft (CABG).

DETAILED DESCRIPTION:
Coronary artery disease and its complications are the leading cause of death in the western world. Diabetes mellitus (DM) is one of the major risk factors to develop coronary artery disease, myocardial infarction and post-infarction complication1-3. Furthermore, mortality from myocardial infarction is almost doubled in diabetic patients compared to non-diabetics4. Despite significant amount of research, the basis for these differences in outcome still remains unclear. The survival of myocardial tissue subjected to ischemia can be increased by the ability to promote growth of new blood vessels into ischemic areas, thus limiting regions of impairment and ultimately preserving myocardial function. Hypoxia inducible factor (HIF) -1 is a transcription factor that promotes the expression of several genes that confer protection against hypoxia/ischemia through angiogenesis, erythropoiesis, vasodilation, and altered glucose metabolism5,6. Our hypothesis is that angiogenesis may be impaired in diabetes mainly via decreased protein expression and activation of HIF-1 and its main downstream target vascular endothelial growth factor (VEGF), as well as the inhibitor angiogenesis factor, angiostatin7, in the heart. Therefore the purpose of this study is to examine whether the angiogenic process during coronary ischemia is influenced by diabetes. To address these questions, HIF-1, VEGF and angiostatin protein expression will be evaluated in atrial tissue obtained from patients with and without diabetes who will undergo coronary bypass surgery. In addition comparison between emergency and elective procedure will be performed in regard to HIF-1 and VEGF protein levels and correlation with chronic statin therapy will be performed.

During the cannulation process, prior to initiation of cardiopulmonary bypass (CPB) during heart surgery, a small piece of the right atrium is cut in order to insert a venous cannula into that chamber. The investigators intend to use this piece of tissue (that is routinely wasted) in our protein and histological analyses.

ELIGIBILITY:
Inclusion Criteria:

1. on-pump CABG
2. 18 years of age & older
3. informed consent

Exclusion Criteria:

1. active malignancy
2. severe lung disease (requiring home O2 therapy)
3. severe anemia<8g/dl
4. patient with moderate or severe renal dysfunction
5. off- pump CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic & non-diabetic CABG patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
tissue levels of HIF-1, VEGF and angiostatin | initiation of CPB/ day 1
  The investigators will evaluate tissue levels of HIF-1, VEGF and angiostatin in diabetic and non-diabetic patients coming for on-pump CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Raphael, MD, Principal Investigator — UVA Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar D, Solomon SD, Kober L, Rouleau JL, Skali H, McMurray JJ, Francis GS, Henis M, O'Connor CM, Diaz R, Belenkov YN, Varshavsky S, Leimberger JD, Velazquez EJ, Califf RM, Pfeffer MA. Newly diagnosed and previously known diabetes mellitus and 1-year outcomes of acute myocardial infarction: the VALsartan In Acute myocardial iNfarcTion (VALIANT) trial. Circulation. 2004 Sep 21;110(12):1572-8. doi: 10.1161/01.CIR.0000142047.28024.F2. Epub 2004 Sep 13. PMID 15364810
- [Background] Zairis MN, Lyras AG, Makrygiannis SS, Psarogianni PK, Adamopoulou EN, Handanis SM, Papantonakos A, Argyrakis SK, Prekates AA, Foussas SG. Type 2 diabetes and intravenous thrombolysis outcome in the setting of ST elevation myocardial infarction. Diabetes Care. 2004 Apr;27(4):967-71. doi: 10.2337/diacare.27.4.967. PMID 15047657
- [Background] Donahoe SM, Stewart GC, McCabe CH, Mohanavelu S, Murphy SA, Cannon CP, Antman EM. Diabetes and mortality following acute coronary syndromes. JAMA. 2007 Aug 15;298(7):765-75. doi: 10.1001/jama.298.7.765. PMID 17699010
- [Background] Abbott RD, Donahue RP, Kannel WB, Wilson PW. The impact of diabetes on survival following myocardial infarction in men vs women. The Framingham Study. JAMA. 1988 Dec 16;260(23):3456-60. PMID 2974889
- [Background] Semenza GL. Hypoxia-inducible factor 1 and the molecular physiology of oxygen homeostasis. J Lab Clin Med. 1998 Mar;131(3):207-14. doi: 10.1016/s0022-2143(98)90091-9. No abstract available. PMID 9523843
- [Background] Semenza GL, Roth PH, Fang HM, Wang GL. Transcriptional regulation of genes encoding glycolytic enzymes by hypoxia-inducible factor 1. J Biol Chem. 1994 Sep 23;269(38):23757-63. PMID 8089148
- [Background] Weihrauch D, Lohr NL, Mraovic B, Ludwig LM, Chilian WM, Pagel PS, Warltier DC, Kersten JR. Chronic hyperglycemia attenuates coronary collateral development and impairs proliferative properties of myocardial interstitial fluid by production of angiostatin. Circulation. 2004 May 18;109(19):2343-8. doi: 10.1161/01.CIR.0000129225.67353.1F. Epub 2004 May 10. PMID 15136506